CLINICAL TRIAL: NCT00687271
Title: A Multicenter, Randomized, Double-Blind, Placebo- and Active-Controlled Study to Assess the Efficacy, and Tolerability of MK-6213 Co-Administered With Atorvastatin in Patients With Primary Hypercholesterolemia
Brief Title: A Study of MK-6213 Co-Administered With Atorvastatin in Participants With Hypercholesterolemia (MK-6213-006)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 6213-006; 2007_514 (Other: Sponsor Registry Number); 2007-003684-41 (EudraCT Number); MK-6314-006 (Other: Merck Study Number)
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- MK-6213 160 mg + Atorvastatin 20 mg (Experimental): 1 MK-6213 160-mg tablet co-administered orally with 1 Atorvastatin 20-mg tablet once daily for 4 weeks
  Interventions: Drug: MK-6213; Drug: Atorvastatin calcium
- Atorvastatin 20 mg (Active Comparator): 1 Atorvastatin 20-mg tablet co-administered orally with 1 tablet of placebo for MK-6312 once daily for 4 weeks
  Interventions: Drug: Atorvastatin calcium; Drug: Placebo for MK-6312 160 mg
- MK-6213 160 mg (Experimental): 1 MK-6213 160-mg tablet co-administered orally with 1 tablet of placebo for Atorvastatin 20-mg once daily for 4 weeks
  Interventions: Drug: MK-6213; Drug: Placebo for Atorvastatin 20 mg
- Placebo (Placebo Comparator): 1 tablet of placebo for MK-6213 160 mg co-administered orally with 1 tablet of placebo for Atorvastatin 20-mg tablet once daily for 4 weeks
  Interventions: Drug: Placebo for MK-6312 160 mg; Drug: Placebo for Atorvastatin 20 mg

INTERVENTIONS:
Drug: MK-6213 — MK-6213 160 mg for 4 weeks.
  Arms: MK-6213 160 mg; MK-6213 160 mg + Atorvastatin 20 mg
Drug: Atorvastatin calcium — atorvastatin calcium 20mg for 4 weeks.
  Other Names: atorvastatin; LIPITOR ®
  Arms: Atorvastatin 20 mg; MK-6213 160 mg + Atorvastatin 20 mg
Drug: Placebo for MK-6312 160 mg
  Arms: Atorvastatin 20 mg; Placebo
Drug: Placebo for Atorvastatin 20 mg
  Arms: MK-6213 160 mg; Placebo

SUMMARY:
The purpose of this study is to test the safety and effectiveness of MK-6213 as compared to MK-6213/Atorvastatin in participants 18 to 75 years) with high cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age at the time of the study with high cholesterol
* Can have diabetes mellitus but is not currently on lipid lowering therapy
* Have a stable weight for >6 weeks

Exclusion Criteria:

* Has significant cardiovascular (heart), renal (kidney), neurologic (nervous system), respiratory (lung), hepatic (liver) or metabolic disease
* history of mental instability or drug/alcohol abuse within the past 5 years
* Pregnant or nursing; human immunodeficiency virus (HIV) positive; history of cancer within the past 5 years or participation in an investigational trial within the last 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2008-06-14 (Actual); Primary Completion 2009-01-08 (Actual); Study Completion 2009-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MK-6213 160 mg + Atorvastatin 20 mg | Atorvastatin 20 mg | MK-6213 160 mg | Placebo
Started | 94 | 96 | 96 | 48
Treated | 94 | 95 | 96 | 48
Completed | 91 | 90 | 91 | 48
Not Completed | 3 | 6 | 5 | 0
Not completed — Adverse Event | 1 | 3 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-6213 160 mg + Atorvastatin 20 mg | Atorvastatin 20 mg | MK-6213 160 mg | Placebo | Total
Number analyzed (Participants) | 94 | 96 | 96 | 48 | 334
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.9 (10.9) | 53.6 (10.2) | 56.2 (10.0) | 54.7 (10.7) | 54.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 60 | 47 | 26 | 178
  Male | 49 | 36 | 49 | 22 | 156

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Blood collected at baseline (predose) and after 4 weeks of treatment to determine LDL-C levels. LDL-C was calculated using the Friedewald equation. If triglycerides (TG) exceeded 400 mg/dL (4.6 mmol/L), LDL-C was determined by reflex beta-quantitation method. The percentage change from baseline at Week 4 was summarized.
Time Frame: Baseline (predose) and Week 4
Population: All participants that received at least 1 dose of study drug, had baseline value for parameter and had data available for timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | MK-6213 160 mg + Atorvastatin 20 mg | Atorvastatin 20 mg | MK-6213 160 mg | Placebo
Number analyzed (Participants) | 92 | 89 | 92 | 47
Percentage Change | -50.7 [-53.8 to -47.5] | -40.6 [-43.8 to -37.4] | -13.3 [-16.5 to -0.1] | 4.6 [0.2 to 9.1]
Statistical Analysis 1: Comparison: MK-6213 160 mg + Atorvastatin 20 mg vs Atorvastatin 20 mg; Test type: Other; Longitudinal Data Analysis (LDA) model; LDA model includes factors for time, treatment, baseline triglyceride (TG) category, and time-by treatment interactions; Difference in Percentage Change = -10.0, 95% CI 2-sided [-14.6 to -5.5]
Statistical Analysis 2: Comparison: MK-6213 160 mg vs Placebo; Test type: Other; LDA model; LDA model includes factors for time, treatment, baseline triglyceride (TG) category, and time-by treatment interactions; Difference in Percentage Change = -17.9, 95% CI 2-sided [-23.4 to -12.5]

2. Secondary Outcome: Percentage of Participants Who Experience at Least 1 Adverse Event (AE)
Description: An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless of whether or not it was considered related to the medicinal product. The percentage of participants that reported at least 1 AE was summarized
Time Frame: Up to 14 days post last dose of study drug (up to 6 weeks)
Population: All participants that received at least 1 dose for study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-6213 160 mg + Atorvastatin 20 mg | Atorvastatin 20 mg | MK-6213 160 mg | Placebo
Number analyzed (Participants) | 94 | 95 | 96 | 48
Percentage of Participants | 33.0 | 37.9 | 29.2 | 41.7

3. Secondary Outcome: Percentage of Participants That Had Study Drug Discontinued Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless of whether or not it was considered related to the medicinal product. The percentage of participants who had study drug discontinued due to an AE was summarized.
Time Frame: up to 4 weeks
Population: All participants that received at least 1 dose for study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-6213 160 mg + Atorvastatin 20 mg | Atorvastatin 20 mg | MK-6213 160 mg | Placebo
Number analyzed (Participants) | 94 | 95 | 96 | 48
Percentage of Participants | 1.1 | 3.1 | 1.0 | 0.0

4. Secondary Outcome: Percentage Change From Baseline in Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C)
Description: Blood collected at baseline (predose) and after 4 weeks of treatment to determine non-HDL-C levels. The percentage change from baseline at Week 4 was summarized.
Time Frame: Baseline (predose) and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | MK-6213 160 mg + Atorvastatin 20 mg | Atorvastatin 20 mg | MK-6213 160 mg | Placebo
Number analyzed (Participants) | 92 | 89 | 92 | 47
Percentage Change | -46.6 [-49.5 to -43.6] | -38.0 [-41.0 to -35.0] | -11.4 [-14.3 to -8.5] | 2.5 [-1.6 to 6.6]
Statistical Analysis 1: Comparison: MK-6213 160 mg + Atorvastatin 20 mg vs Atorvastatin 20 mg; Test type: Other; LDA model; LDA model includes factors for time, treatment, baseline triglyceride (TG) category, and time-by treatment interactions; Difference in Percentage Change = -8.6, 95% CI 2-sided [-12.7 to -4.4]
Statistical Analysis 2: Comparison: MK-6213 160 mg vs Placebo; Test type: Other; LDA model; LDA model includes factors for time, treatment, baseline triglyceride (TG) category, and time-by treatment interactions; Diffence in Percentage Change = -13.9, 95% CI 2-sided [-18.9 to -8.9]

5. Secondary Outcome: Percentage Change From Baseline in Apolipoprotein B (ApoB)
Description: Blood collected at baseline (predose) and after 4 weeks of treatment to determine ApoB levels. The percentage change from baseline at Week 4 was summarized.
Time Frame: Baseline (predose) and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | MK-6213 160 mg + Atorvastatin 20 mg | Atorvastatin 20 mg | MK-6213 160 mg | Placebo
Number analyzed (Participants) | 92 | 89 | 92 | 47
Percentage Change | -40.4 [-43.1 to -37.7] | -32.7 [-35.4 to -30.0] | -8.8 [-11.5 to -6.1] | 3.5 [-0.3 to 7.2]
Statistical Analysis 1: Comparison: MK-6213 160 mg + Atorvastatin 20 mg vs Atorvastatin 20 mg; Test type: Other; LDA model; LDA model includes factors for time, treatment, baseline triglyceride (TG) category, and time-by treatment interactions; Difference in Percentage Change = -7.7, 95% CI 2-sided [-11.5 to -3.9]
Statistical Analysis 2: Comparison: MK-6213 160 mg vs Placebo; Test type: Other; LDA model; LDA model includes factors for time, treatment, baseline triglyceride (TG) category, and time-by treatment interactions; Difference in Percentage Change = -12.2, 95% CI 2-sided [-16.8 to -7.6]

6. Secondary Outcome: Percentage Change From Baseline in Total Cholesterol (TC)
Description: Blood collected at baseline (predose) and after 4 weeks of treatment to determine TC levels. The percentage change from baseline at Week 4 was summarized.
Time Frame: Baseline (predose) and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | MK-6213 160 mg + Atorvastatin 20 mg | Atorvastatin 20 mg | MK-6213 160 mg | Placebo
Number analyzed (Participants) | 92 | 89 | 92 | 47
Percentage Change | -35.1 [-37.4 to -32.7] | -27.6 [-30.0 to -25.2] | -8.5 [-10.9 to -6.2] | 2.5 [-0.8 to 5.8]
Statistical Analysis 1: Comparison: MK-6213 160 mg + Atorvastatin 20 mg vs Atorvastatin 20 mg; Test type: Other; LDA model; LDA model includes factors for time, treatment, baseline triglyceride (TG) category, and time-by treatment interactions; Difference in Percentage Change = -7.4, 95% CI 2-sided [-10.8 to -4.1]
Statistical Analysis 2: Comparison: MK-6213 160 mg vs Placebo; Test type: Other; LDA model; LDA model includes factors for time, treatment, baseline triglyceride (TG) category, and time-by treatment interactions; Difference in Percentage Change = -11.0, 95% CI 2-sided [-15.1 to -7.0]

7. Secondary Outcome: Percentage Change From Baseline in HDL-C
Description: Blood collected at baseline (predose) and after 4 weeks of treatment to determine HDL-C levels. The percentage change from baseline at Week 4 was summarized.
Time Frame: Baseline (predose) and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | MK-6213 160 mg + Atorvastatin 20 mg | Atorvastatin 20 mg | MK-6213 160 mg | Placebo
Number analyzed (Participants) | 92 | 89 | 92 | 47
Percentage Change | 3.8 [0.9 to 6.8] | 6.2 [3.2 to 9.2] | 1.4 [-1.6 to 4.3] | 2.1 [-2.1 to 6.2]
Statistical Analysis 1: Comparison: MK-6213 160 mg + Atorvastatin 20 mg vs Atorvastatin 20 mg; Test type: Other; LDA model; LDA model includes factors for time, treatment, baseline triglyceride (TG) category, and time-by treatment interactions; Dfferecne in Percentage Change = -2.4, 95% CI 2-sided [-6.6 to 1.8]
Statistical Analysis 2: Comparison: MK-6213 160 mg vs Placebo; Test type: Other; LDA model; LDA model includes factors for time, treatment, baseline triglyceride (TG) category, and time-by treatment interactions; Difference in Percentage Change = -0.7, 95% CI 2-sided [-5.8 to 4.4]

8. Secondary Outcome: Percentage Change From Baseline in TG
Description: Blood collected at baseline (predose) and after 4 weeks of treatment to determine TG levels. The percentage change from baseline at Week 4 was summarized.
Time Frame: Baseline (predose) and Week 4
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-6213 160 mg + Atorvastatin 20 mg | Atorvastatin 20 mg | MK-6213 160 mg | Placebo
Number analyzed (Participants) | 92 | 89 | 92 | 47
Percentage of Participants | -24.2 [-29.6 to -18.9] | -25.9 [-32.1 to -19.7] | 1.6 [-6.9 to 10.1] | -7.1 [-17.2 to 3.0]
Statistical Analysis 1: Comparison: MK-6213 160 mg + Atorvastatin 20 mg vs Atorvastatin 20 mg; Test type: Other; LDA model; LDA model includes factors for time, treatment, baseline triglyceride (TG) category, and time-by treatment interactions; Difference in Percentage Change = -1.0, 95% CI 2-sided [-7.7 to 5.9]
Statistical Analysis 2: Comparison: MK-6213 160 mg vs Placebo; Test type: Other; LDA model; LDA model includes factors for time, treatment, baseline triglyceride (TG) category, and time-by treatment interactions; Difference in Percentage Change = 5.5, 95% CI 2-sided [-4.6 to 16.9]

ADVERSE EVENTS:
Time Frame: up to 2 weeks post last dose (up to 6 weeks total)
Description: Population included all participants that received at least 1 dose of study drug.
Arm/Group | MK-6213 160 mg + Atorvastatin 20 mg | Atorvastatin 20 mg | MK-6213 160 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/95 | 0/96 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/95 | 0/96 | 0/48
Other Adverse Events (participants affected / at risk) | 3/94 | 5/95 | 5/96 | 2/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-6213 160 mg + Atorvastatin 20 mg (N=94) | Atorvastatin 20 mg (N=95) | MK-6213 160 mg (N=96) | Placebo (N=48)
Headache (Nervous system disorders) | 3 (3) | 5 (7) | 5 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines